CLINICAL TRIAL: NCT05328648
Title: Randomized Controlled Trial to Address Unintended Pregnancy Rates in Low Resource Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Safe Water and AIDS Project (Other); Innovations for Poverty Action (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-2217; 1R01HD101453-01A1 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-05

CONDITIONS: Contraceptive Usage; Unintended Pregnancy
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community Score Card (Experimental): In the Community Score Card approach, community members come together to document challenges they encounter when seeking services and develop a corresponding set of indicators that can be used to produce a validated facility score. The score is shared with the community and a collaborative process between key community members and facility staff takes place to develop feasible solutions and a strategic action plan.
  Interventions: Behavioral: Community Score Card
- Citizen Report Card (Experimental): In the Citizen Report Card approach, individual-level feedback is collected from actual clients of target facilities, via a structured questionnaire, to assess facility performance and generate a public record of service quality. In addition to sharing the final report card with communities, engaged policymakers are invited to use the citizen feedback to improve service delivery.
  Interventions: Behavioral: Citizen Report Card
- Control (No Intervention): Communities in the control arm will not receive an intervention.

INTERVENTIONS:
Behavioral: Community Score Card — In Community Score Card intervention, all communities associated with the targeted facilities will assess the primary barriers to quality family planning service delivery and develop indicators. The communities will then each complete the score card and generate ideas for quality improvement. Family planning providers in the target facilities will meet and determine the barriers to high quality family planning service delivery. Providers will decide on priority areas and make suggestions for improving service delivery. Study facilitators will bring these two groups together to share their respective score cards and jointly develop an action. Within the action plan, agreed upon responsibilities will be assigned and a timeline will be communicated.
  Arms: Community Score Card
Behavioral: Citizen Report Card — Citizen Report Card (CRC): The data from the CRC questionnaire will be analyzed and translated into a report card. Extensive dissemination activities will ensure the CRC is widely shared with members of the community. The goal is to create a public record of service quality.
  Arms: Citizen Report Card

SUMMARY:
This is a clinical trial investigating the impact of social accountability interventions on contraceptive use in Western Kenya. Social accountability interventions aim to improve the performance of healthcare providers via public monitoring of provider performance. This study aims to implement and evaluate two social accountability interventions: the community score card and the citizen report card. All public-sector healthcare facilities in Kisumu Country will be considered for enrollment; facility staff and residents of corresponding facility catchment areas will be randomized to one of the two treatments or the control arm.

DETAILED DESCRIPTION:
Purpose: The primary objective is to examine the health impact of implementing social accountability interventions in communities served by public-sector healthcare facilities in Western Kenya. The first aim is to assess the impact of two social accountability approaches on contraceptive use. The second aim is to assess the impact of these approaches on community empowerment, agency, and quality of care. Third third aim is to assess the scalability of these approaches to additional settings. The study will be carried out in Kisumu county, Kenya. This study design is a three-arm cluster-randomized controlled experiment in which all public healthcare facilities in the county will be randomized to one of three study arms: 1. Community Score Card treatment, 2. Citizen Report Card treatment or 3. control.

Before and after implementing the two treatments, individual- and facility-level pre- and postintervention surveys will be conducted.

The individual-level surveys will be conducted within a representative sample of women of reproductive age (ages 18 to 49), stratified by study arm and cluster, and will be used to establish the primary outcome, modern contraceptive use, in all three study arms, pre- and post-treatment. The individual-level surveys will also measure multiple linking constructs such as community empowerment and quality of care.

The facility-level surveys will be conducted in a census of all public-sector facilities located in Kisumu county and will be used to measure quality of family planning service delivery and negative provider behaviors such as informal payments, provider absenteeism, and client mistreatment. For the facility-level surveys, family planning service quality and negative provider behaviors will be measured via interviews with one to ten providers, depending on total staff at each of the facilities. This will result in approximately 385 provider interviews, with approximately 128 in each study arm. Unannounced visitors and mystery clients will also be deployed to secure less biased estimates of provider absenteeism, informal fee solicitation, and disrespectful/biased treatment of clients; mystery clients will also collect data on traditional measures of family planning service quality such as choice of methods and information on side effects. All facilities in Kisumu will receive two unannounced visits and three mystery client visits.

Post-treatment, the individual-level survey will be repeated, within a newly sampled cross-section of the population. All facility-level data collection in all public facilities in the county will also be repeated. The changes in contraceptive use, quality of care, and community engagement resulting from the Community Score Card and the Citizen Report Card interventions will be evaluated via data collected in these pre- and post-intervention surveys.

Following the interventions, four focus groups (two/arm) will be conducted with key facilitators in the two intervention approaches to better understand implementation challenges and potential barriers to scaling up these interventions to other regions or countries. In-depth interviews will be undertaken with health care providers and community members to assess the potential for scale-up of these interventions. Interviews with 30 providers and community members will be completed in each of the two intervention arms (15/arm). Respondents will be asked to reflect on their experiences with the intervention and provide feedback for areas for improvement and scalability.

The Interventions

The Community Score Card Approach (CSC) CSC Summary: In the Community Score Card approach, community members come together to document challenges they encounter when seeking services and develop a corresponding set of indicators that can be used to produce a validated facility score. The score is shared with the community and a collaborative process between key community members and facility staff takes place to develop feasible solutions and a strategic action plan.

CSC Procedures:

Step 1: Preparation. The communities and facility staff will be engaged and sensitized to the community score card via a meeting that discusses the community score card purpose and approach; a date, location, and general process for conducting the CSCs will be selected/designed.

Step 2: Conducting the CSC with target communities. During this phase, all communities associated with the targeted facilities will assess the primary barriers to quality family planning service delivery and develop corresponding indicators, assisted by an experienced facilitator. The communities will then each complete the score card and generate ideas for quality improvement.

Step 3: Conducting the CSC with family planning providers. Family planning providers in the target facilities will meet and determine the barriers to high quality family planning service delivery. Providers will decide on priority areas and make suggestions for improving service delivery. Providers may derive a similar list of issues/indicators as the community.

Step 4: Connecting the patients and providers and determining an action plan. Family planning patients and providers - as well as community leaders and process facilitators - will come together to present their findings and to jointly determine the priority areas and develop an action plan. Within the action plan, agreed upon responsibilities will be assigned and a timeline will be communicated.

Step 5: Implementing the action plan and continuous monitoring. In this final stage, the action plan will be carried out over a period of approximately six months, with community members and service providers in charge of monitoring implementation and progress. After a period of six months, the patient and provider score cards will be repeated.

The Citizen Report Card Approach (CRC) CRC Summary: In this approach, individual-level feedback is collected from actual clients of target facilities, via a structured questionnaire, to assess facility performance and generate a public record of service quality. In addition to sharing the final report card with communities, engaged policymakers are invited to use the citizen feedback to improve service delivery.

Step 1: Preparing for data collection and dissemination. The PI will consult with the Kisumu County Health Director to confirm the geographic coverage of the citizen report card. The PI will also collaborate with staff in the county health office to develop a post-survey publicity strategy. The strategy could include community dialogues, radio call-in shows, television, and newspaper coverage.

Step 2: Designing the CRC survey. As part of the intervention, three focus groups will be conducted (two with family planning clients stratified into younger versus older women and one with service providers). This will help to identify key service challenges and inform the content of the CRC questionnaire by allowing citizens to articulate and prioritize relevant indicators for monitoring and reporting on service provider performance. Focus groups with service providers may elicit suggestions for the type of feedback they would find most useful for improving their service delivery. In general, both providers and clients will be asked about the problem areas related to family planning service delivery. Once focus group discussions are completed and the data are analyzed, investigators will identify the prominent themes related to family planning service delivery that emerge from the focus group data. In turn, these themes will inform the main content of the CRC questionnaire.

Step 4: Analyze the data. Data from the CRC questionnaire will be analyzed and results will be translated into a report card. The report card will also be translated into the local languages (Kiswahili and Dholuo) so that it is accessible to a broad range of stakeholders.

Step 5: Disseminate results to the community. Extensive dissemination activities will ensure the Citizen Report Card is widely shared with members of the community. Report card findings will be presented at a high-profile press conference and press kit materials with short, readable stories will be distributed to members of the print, radio, and television media. The goal is to create a public record of service quality.

ELIGIBILITY:
Inclusion Criteria:

Women's level survey:

* Women aged 18-49 years;
* Reside in randomly selected households.

Provider Survey:

* Healthcare service provider;
* Provides family planning or reproductive health services;
* Works in a public-sector healthcare facility located in Kisumu County.

Focus Group Discussions:

* Key intervention facilitators;
* Over the age of 18 years

Qualitative In-Depth Interviews:

* Community members in Kisumu County who participated in intervention activities;
* Family planning service providers who work within a public-sector healthcare facility in Kisumu County;
* Over 18 years of age.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants are eligible if they self-identify as female.
Enrollment: 5726 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Tumlinson, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Innovations for Poverty Action, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
The study will make available its data after it's been de-identified. These will be shared with researchers who provide a methodologically sound proposal to the study team. Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose will then receive the requested data. Proposals should be directed to Katherine Tumlinson, PhD at ktumlin@email.unc.edu. To gain access, data requestors will need to sign a data use agreement.
Supporting Information: Study Protocol
Time Frame: Data will be made available beginning 9 months and ending 36 months after article publication.
Access Criteria: Ethics approval and executed data use agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two types of participants were enrolled at two time points. 2484 and 2501 women were enrolled in the individual-level survey at baseline and endline, respectively. 345 and 396 healthcare providers (staff) were enrolled in the facility-level survey at baseline and endline, respectively. The facility-level surveys were conducted across 137 public-sector facilities (i.e., the unit of randomization). 2484+345+2501+396 = 5,726. No facility facilitators were enrolled.
Pre-assignment Details: All public health facilities in the study area were included and randomly assigned to 1 of 3 intervention arms. Data was collected through 2 cross-sectional surveys, at baseline and 12 months following intervention implementation. A random sample of reproductive age women and up to 10 providers at each facility, were surveyed at both time points. The sum of participants represents the total number of interviews not the individual respondents, as participants could be sampled at both time points.
Units Other Than Participants: Facilities
Period: Baseline Women
Arm/Group | Community Score Card | Citizen Report Card | Control
Started (Reflects women surveyed at Baseline.) | 828; 45 Facilities | 835; 46 Facilities | 821; 46 Facilities
Completed | 828; 45 Facilities | 835; 46 Facilities | 821; 46 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities
Period: Baseline Providers
Arm/Group | Community Score Card | Citizen Report Card | Control
Started | 106; 45 Facilities | 133; 46 Facilities | 106; 46 Facilities
Providers Interviewed (Reflects providers surveyed at Baseline.) | 106; 45 Facilities | 133; 46 Facilities | 106; 46 Facilities
Providers Not Interviewed (Providers who were either too busy or could not be found to participate in interview. However, their attendance was taken although they were not enrolled.) | 23; 17 Facilities | 18; 13 Facilities | 28; 15 Facilities
Completed | 106; 45 Facilities | 133; 46 Facilities | 106; 46 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities
Period: Endline Women
Arm/Group | Community Score Card | Citizen Report Card | Control
Started (Reflects women surveyed at Endline.) | 822; 45 Facilities | 850; 46 Facilities | 829; 46 Facilities
Completed | 822; 45 Facilities | 850; 46 Facilities | 829; 46 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities
Period: Endline Providers
Arm/Group | Community Score Card | Citizen Report Card | Control
Started | 148; 45 Facilities | 125; 46 Facilities | 123; 46 Facilities
Providers Interviewed (Reflects providers surveyed at Endline.) | 148; 45 Facilities | 125; 46 Facilities | 123; 46 Facilities
Providers Not Interviewed (Providers who were either too busy or could not be found to participate in interview. However, their attendance was taken although they were not enrolled.) | 6; 5 Facilities | 6; 6 Facilities | 6; 5 Facilities
Completed | 148; 45 Facilities | 125; 46 Facilities | 123; 46 Facilities
Not Completed | 0; 0 Facilities | 0; 0 Facilities | 0; 0 Facilities

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Score Card | Citizen Report Card | Control | Total
Number analyzed (Participants) | 1904 | 1943 | 1879 | 5726
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics are summarized by the number of participants completing each survey period.
  years
    Baseline Women: number analyzed (Participants) | 828 | 835 | 821 | 2484
    Baseline Women | 30.43 (8.44) | 30.99 (8.57) | 30.22 (8.72) | 30.55 (8.58)
    Baseline Providers: number analyzed (Participants) | 106 | 133 | 106 | 345
    Baseline Providers | 36.25 (7.82) | 37.52 (8.83) | 37.96 (8.54) | 37.26 (8.45)
    Endline Women: number analyzed (Participants) | 822 | 850 | 829 | 2501
    Endline Women | 30.66 (8.36) | 31.31 (8.49) | 31.11 (8.52) | 31.03 (8.46)
    Endline Providers: number analyzed (Participants) | 148 | 125 | 123 | 396
    Endline Providers | 38.05 (7.73) | 39.52 (8.22) | 38.93 (8.55) | 38.79 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics are summarized by the number of participants completing each survey period.
  Participants
    Baseline Women: number analyzed (Participants) | 828 | 835 | 821 | 2484
    Baseline Women: Female | 828 | 835 | 821 | 2484
    Baseline Women: Male | 0 | 0 | 0 | 0
    Baseline Providers: number analyzed (Participants) | 106 | 133 | 106 | 345
    Baseline Providers: Female | 69 | 100 | 84 | 253
    Baseline Providers: Male | 37 | 33 | 22 | 92
    Endline Women: number analyzed (Participants) | 822 | 850 | 829 | 2501
    Endline Women: Female | 822 | 850 | 829 | 2501
    Endline Women: Male | 0 | 0 | 0 | 0
    Endline Providers: number analyzed (Participants) | 148 | 125 | 123 | 396
    Endline Providers: Female | 100 | 90 | 99 | 289
    Endline Providers: Male | 48 | 35 | 24 | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 1904 | 1943 | 1879 | 5726

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Current Modern Contraceptive Use
Description: The measure of current modern contraceptive use is a binary variable (0=non-use; 1=use), attained by first asking participants, "Are you (or your partner) currently doing something or using any method to delay or avoid getting pregnant?" Those with an affirmative response are then asked, "What method are you using?" Modern contraceptive methods will be defined to include female or male sterilization, intrauterine device, implant, injectable contraception, oral contraceptive pill, male or female condom, and any other modern methods. The percent of women using modern contraceptives at baseline was subtracted from the percent using modern contraceptives at endline, and that difference is reported.
Time Frame: Baseline, 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
percentage of participants | -1.1 | 1.4 | 1.5

2. Primary Outcome: Mean Knowledge of Patient Rights Score
Description: The measure of women's knowledge of patient rights is a 7 item scale with answers on a 5 point Likert scale. Possible scores range from 7 to 35. Higher scores reflect greater knowledge of patient rights. The measure of women's knowledge of patient rights is implemented in the women's individual-level questionnaire in the pre- and post-intervention surveys. The percent change in the mean score across all women is presented, using the formula (endline-baseline)/baseline.
Time Frame: Baseline, at the end of 12-month intervention (Endline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
score on a scale
  Baseline | 18.1 (3.7) | 18.0 (3.6) | 18.0 (3.6)
  Endline | 18.0 (3.8) | 17.5 (3.6) | 17.8 (3.6)

3. Primary Outcome: Mean Women's Agency Within Their Community Score
Description: The measure of women's agency within their community is an 8 item scale. Answers are on a 5 point scale with options "Completely sure" "Sure" "Neither sure or unsure" "Not sure" or "Not sure at all." Possible scores range from 8 to 40. Higher scores reflect greater agency for women within their community. The measure of women's agency within their community is implemented in the women's individual-level questionnaire in the pre- and post-intervention surveys.
Time Frame: Baseline, at the end of 12-month intervention (Endline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
score on a scale
  Baseline | 20.8 (6.5) | 21.1 (6.4) | 21.2 (6.1)
  Endline | 21.5 (6.7) | 21.2 (7.2) | 21.7 (7.1)

4. Primary Outcome: Mean Women's Agency Within a Healthcare Facility
Description: The measure of women's agency within a healthcare facility is a 2 item scale. Answers are on a 5 point scale with options "Completely sure" "Sure" "Neither sure or unsure" "Not sure" or "Not sure at all." Possible scores range from 2 to 10. Higher scores reflect greater agency for women within a healthcare facility. The measure of women's agency within a healthcare facility is implemented in the women's individual-level questionnaire in the pre- and post-intervention surveys.
Time Frame: Baseline, at the end of 12-month intervention (Endline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
score on a scale
  Baseline | 5.8 (2.1) | 6.0 (2.0) | 5.9 (2.2)
  Endline | 5.6 (2.1) | 5.7 (2.2) | 5.8 (2.0)

5. Primary Outcome: Mean Women's Facility Satisfaction Score
Description: The measure of women's facility satisfaction is an 11 item scale with answers on a 5 point Likert scale. Possible scores range from 11 to 55. Higher scores reflect greater facility satisfaction. The measure of women's facility satisfaction is implemented in the women's individual-level questionnaire in the pre- and post-intervention surveys.
Time Frame: Baseline, at the end of 12-month intervention (Endline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
score on a scale
  Baseline | 23.6 (4.2) | 23.1 (4.0) | 23.2 (4.1)
  Endline | 22.4 (4.4) | 22.5 (4.7) | 23.0 (4.3)

6. Primary Outcome: Mean Community Empowerment Score
Description: The measure of community empowerment is a 4 item scale with answers on a 5 point Likert scale. Possible scores range from 4 to 20. Higher scores reflect greater community empowerment. The measure of community empowerment is implemented in the women's individual-level questionnaire in the pre- and post-intervention surveys.
Time Frame: Baseline, at the end of 12-month intervention (Endline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
score on a scale
  Baseline | 9.9 (3.9) | 10.0 (3.8) | 10.4 (4.1)
  Endline | 9.8 (4.1) | 10.0 (4.5) | 10.0 (4.1)

7. Primary Outcome: Mean Community Involvement
Description: There are three indicators measuring community involvement: In the last 12 months, have you
  1. been an active member in any organized group in your community, for example a women's group, a religious group, or other community group?
  2. received help from any organized group in your community, for example a women's group, a religious group, or other community group? Help could include emotional support, economic assistance, or helping you to learn or do things.
  3. joined together with other people in your community to improve health services for women or children?
  All indicators have a binary response option (Yes/No). A value of 1 was assigned to all affirmative responses and created a scale (0-3). Higher scores reflect more community involvement.
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
score on a scale
  Baseline | 1.3 (1.1) | 1.3 (1.1) | 1.3 (1.1)
  Endline | 1.4 (1.0) | 1.4 (1.0) | 1.4 (1.1)

8. Primary Outcome: Mean Perceived Quality of Family Planning Service Delivery Score
Description: Perceived quality of family planning service delivery is measured via 20 survey questions with different answer options, ranging from binary to four response options. All but two of the 20 variables were binary yes/no (0/1) response options; the remaining two variables were initially variables with four response options that were collapsed to binary response options (0/1). Possible scores range from 0 to 20. Higher scores reflect greater perceived quality of family planning service delivery. The measure of perceived quality is implemented in the women's individual-level questionnaire in the pre- and post-intervention surveys.
Time Frame: Baseline, at the end of 12-month intervention (Endline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 1650 | 1685 | 1650
score on a scale
  Baseline | 17.3 (2.3) | 17.4 (2.2) | 17.3 (2.6)
  Endline | 17.0 (2.6) | 17.1 (2.5) | 17.1 (2.5)

9. Primary Outcome: Percent Change in Provider Absenteeism
Description: The measure of absenteeism is a binary variable obtained using a roster of healthcare providers to assess provider absence. Response options for each provider include Yes and No and up to 10 providers at each facility will be assessed for absence. The percent of providers absent will be measured by taking the number of providers absent and dividing by the total number of providers listed on the roster. The percent change in absenteeism is calculated by subtracting the baseline from the endline and dividing by the baseline. The measure of provider absenteeism is implemented in the facility-level unannounced visitor questionnaire in the pre- and post-intervention surveys. Enumerators took attendance, using a pre-obtained roster of all scheduled healthcare providers, on the day of data collection. Not all healthcare providers were enrolled/interviewed. No non-provider staff were enrolled.
Time Frame: Baseline, 12 months
Measure: Number; unit: percent change in providers absent
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 283 | 282 | 263
percent change in providers absent | -5.9 | 15.2 | -8.3

10. Primary Outcome: Percent Change in the Number of Mystery Client Observations of Providers in Which the Mystery Client Answered in the Affirmative to the Full Method Information Index Plus (MII+)
Description: The Method Information Index Plus (MII+) consists of four indicators: "Were you informed about other methods?" "Were you informed about side effects?" "Were you told what to do if you experienced side effects?" "Were you told about the possibility of switching to another method if the method you selected was not suitable?" The reported value is the percentage of mystery client (MC) observations in which the mystery client answered in the affirmative for all four indicators in the index. The percent change in affirmative observations is calculated by subtracting the baseline from the endline and dividing by the baseline. MII+ is measured in the mystery client observation guide in the pre- and post-intervention surveys. Highly experienced, well-trained data collectors served as mystery clients. These enumerators were part of the study team and not participants who signed informed consent.
Time Frame: Baseline, 12 months
Population: Each facility was observed by 3 different mystery clients at both Baseline and Endline. The 3 observations per facility do not necessarily represent 3 different providers. No identifying information was collected from any provider observed by a mystery client. The Overall Number of Participants shown above reflect mystery client observations.
Measure: Number; unit: percent change
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 270 | 276 | 276
percent change | -22.8 | -67.0 | -64.1

11. Primary Outcome: Percent Change in Mystery Client Observations With Informal Payment Solicitation
Description: The measure of informal payment solicitation is a binary variable obtained by asking mystery clients whether they were asked by facility staff to pay when seeking family planning services at a public-sector healthcare facility. Response options include Yes and No. The percent of mystery client visits in which an informal payment is solicited will be measured by taking the number of mystery client visits for which an informal fee is solicited and dividing by the total number of mystery client visits. The percent change in mystery client observations with informal payment solicitation is calculated by subtracting the baseline from the endline and dividing by the baseline.The measure of informal payments is implemented in the mystery client questionnaire in the pre- and post-intervention surveys. Highly experienced, well-trained data collectors served as mystery clients. These enumerators were part of the study team and not participants who signed informed consent.
Time Frame: Baseline, 12 months
Population: Each facility was observed by 3 different mystery clients at both Baseline and Endline. The 3 observations per facility do not necessarily represent 3 different providers. No identifying information was collected from any provider observed by a mystery client. The Overall Number of Participants shown above reflect mystery client observations of providers.
Measure: Number; unit: percent change
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 270 | 276 | 276
percent change | -34.0 | -20.6 | -25.2

12. Primary Outcome: Percent Change in the Number of Mystery Client Observations Identifying Patient Mistreatment
Description: The measure of patient mistreatment is a binary variable obtained by asking mystery clients "Did your provider do any of the following?" Response options include Shouted at me; Scolded me or treated me with scorn; Threatened to withhold services; Called me by an insulting name; Laughed at me; Other type of disrespect, please explain. If the mystery client selects any of the response options, patient mistreatment is identified. The percent of mystery client visits in which patient mistreatment occurs will be measured by taking the number of mystery client visits for which mistreatment occurs and dividing by the total number of mystery client visits. The measure of patient mistreatment is implemented in the mystery client questionnaire in the pre- and post-intervention surveys. Highly experienced, well-trained data collectors served as mystery clients. These enumerators were part of the study team and not participants who signed informed consent.
Time Frame: Baseline, 12 months
Population: Facilities were observed by 3 different mystery clients at both Baseline and Endline. The 3 observations per facility do not necessarily represent 3 different providers. No identifying information was collected from any provider observed by a MC. The Overall Number of Participants shown above reflect MC observations of providers. The percent change in MC observations with informal payment solicitation is calculated by subtracting the baseline from the endline and dividing by the baseline.
Measure: Number; unit: percent change mistreatment observations
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 270 | 276 | 276
percent change mistreatment observations | 53.2 | 161.9 | 118.4

13. Primary Outcome: Mean Close-to-Community (CTC) Provider Motivation Indicator Score
Description: The CTC provider motivation indicator scale is a 12 item scale. Answers are on a 5 point Likert scale. Possible scores range from 12 to 60. Higher scores reflect greater provider motivation. The measure of provider motivation is implemented in the facility-level provider's questionnaire in the pre- and post-intervention surveys.
Time Frame: Baseline, at the end of 12-month intervention (Endline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Score Card | Citizen Report Card | Control
Number analyzed (Participants) | 254 | 258 | 229
score on a scale
  Baseline | 17.9 (4.3) | 17.4 (4.3) | 18.3 (4.9)
  Endline | 18.4 (4.7) | 18.5 (4.6) | 17.8 (4.5)

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed for the study
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed within the study
Arm/Group | Community Score Card | Citizen Report Card | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT05328648/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT05328648/ICF_000.pdf